CLINICAL TRIAL: NCT04589351
Title: Kidney Fat in Type 2 Diabetes & Diabetic Kidney Disease and the Effects of Ezetimibe: A Cross-Sectional Study and Randomized, Placebo-Controlled Trial
Brief Title: Kidney Fat in Type 2 Diabetes and the Effects of Ezetimibe
Acronym: DiaKidZ
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); Aalborg University Hospital (Other); Capital Region's Pharmacy (Region Hovedstadens Apotek), Marielundvej 25, 2730 Herlev, Denmark (Unknown); Alessia Fornoni, MD PhD, Professor of Medicine, Chief, Katz Family Division of Nephrology and Hypertension (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16032020; 2020-001155-40 (EudraCT Number)
Record Dates: First submitted 2020-10-02; First posted 2020-10-19 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — Ezetimibe

STUDY DESIGN:
Intervention Model Description: This study consists of a cross-sectional study and an intervention trial. The latter is a single-center, randomized, double-blinded, placebo-controlled and parallel trial in participants with T2D and non-severe diabetic kidney disease.
  Trial participants (n=60), by virtue of their baseline examinations (e.g. MR-examinations), also participate in the cross-sectional part of this study where they constitute one of three groups. The other two groups contain controls (n=30) and individuals with T2D and no diabetic kidney disease (n=30).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To ensure blinding to the trial drug, the tablets containing either ezetimibe or placebo are incapsulated with gelatin and thus identical in appearance (size, color and shape).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ezetimibe (Active Comparator): One treatment period of 16 weeks with1 capsule of ezetimibe 10mg per day, as add-on to standard care.
  Interventions: Drug: Ezetimibe 10mg
- Placebo (Placebo Comparator): One treatment period of 16 weeks with 1 capsule of matching placebo per day, as add-on to standard care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ezetimibe 10mg — Ezetimibe is a cholesterol absorption inhibitor with marketing approval. The recommended dose as per label is 10mg once a day.
  Arms: Ezetimibe
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
In this study, we seek to explore the importance of fat accumulation in the kidneys in relation to diabetic kidney disease (DKD). To do this, we conduct an intervention trial in individuals with type 2 diabetes (T2D) and DKD where we investigate whether the inhibition of intestinal cholesterol absorption with ezetimibe affects albuminuria (a strong risk factor for diabetic complications) and kidney fat accumulation. At the same time and to confirm that kidney fat accumulation is, in fact, abnormal in T2D and DKD, we conduct a cross-sectional study in which we compare kidney fat accumulation in participants at baseline from the intervention trial with a group of individuals with T2D and no DKD and a group of healthy individuals.

DETAILED DESCRIPTION:
Objective:

1. To compare cross-sectionally the fractions of kidney lipid between controls, individuals with type 2 diabetes and no diabetic kidney disease and individuals with type 2 diabetes and non-severe diabetic kidney disease.
2. To assess by intervention trial whether ezetimibe reduces albuminuria and kidney parenchymal triglyceride fraction in individuals with type 2 diabetes and non-severe diabetic kidney disease.

Design:

1. Cross-sectional study on 30 controls, 30 individuals with type 2 diabetes and no diabetic kidney disease and 60 individuals with type 2 diabetes and non-severe diabetic kidney disease.
2. Single-center, randomized, double-blinded, placebo-controlled and parallel intervention trial in 60 individuals with type 2 diabetes and non-severe diabetic kidney disease Comparative treatment regime: Ezetimibe 10mg per day versus placebo for 16 weeks

   Primary endpoint in cross-sectional study:
   * Kidney parenchymal triglyceride fraction (estimated by magnetic resonance spectroscopy)

   Primary endpoint in intervention trial:
   * Urinary albumin creatinine ratio

   Secondary endpoint in intervention trial:

   • Kidney parenchymal triglyceride fraction (estimated by magnetic resonance spectroscopy)

   Main eligibility criteria for control group (cross-sectional study alone):

   • Age 40-75 years

   • No diabetes mellitus

   • No kidney disease or urinary albumin creatinine ratio ≥ 30mg/g

   • No contraindication to examination by magnetic resonance

   Main eligibility criteria for group of individuals with type 2 diabetes and no diabetic kidney disease (cross-sectional study alone):

   • Age 40-75 years
   * Type 2 diabetes
   * No kidney disease or urinary albumin creatinine ratio ≥ 30mg/g
   * No contraindication to examination by magnetic resonance

   Main eligibility criteria for group of individuals with type 2 diabetes and non-severe diabetic kidney disease (intervention trial):

   • Age 40-75 years
   * Type 2 diabetes
   * Estimated glomerular filtration rate ≥30ml/min/1,73m2
   * Urinary albumin creatinine ratio ≥ 30mg/g
   * No contraindication to examination by magnetic resonance

   Recruitment
   * Controls are recruited via announcements on relevant websites and, if necessary, in newspapers
   * Individuals with type 2 diabetes are primarily recruited from the ambulatory at Steno Diabetes Center Copenhagen

ELIGIBILITY:
Inclusion criteria for the intervention trial

* Age ≥ 40 and ≤ 75 years
* T2D (World Health Organization criteria)
* eGFR ≥ 30ml/min/1,73m2 at screening
* Persistent UACR ≥ 30mg/g (in more than two out of three valid measurements over a minimum of three months)
* LDL > 1.5mmol/L at screening
* Ability to communicate with the investigator and give informed consent

Exclusion criteria for the intervention trial

* Chronic kidney disease primarily ascribed to other causes than diabetes
* Acute kidney disease within 3 months
* No UACR ≥ 3000mg/g in history
* Current or recent (within 3 months) treatment with ezetimibe
* Initiation or adjustment in dosage within 1 month of an angiotensin-converting enzyme (ACE) inhibitor, angiotensin II receptor blocker (ARB), glucagon-like peptide-1 receptor (GLP-1RA) agonists, sodium-glucose cotransporter 2 (SGLT-2) inhibitors or anti-dyslipidemia drug, e.g. a statin
* Any contraindication to MR-examination (e.g. magnetic foreign body that cannot easily be removed from the body prior to the examination, claustrophobia or body size not compatible with the scanner)
* Intolerance to trial drug components
* Any previous major organ transplantation
* Elective major surgery during the trial
* Pregnancy, planned pregnancy or breastfeeding during the trial
* Insufficient contraception during the trial in women of childbearing potential
* Severe alcohol consumption or abuse of recreational drugs
* Moderate to severe liver failure (Child Pugh 7-15)
* Any surgical or medical condition which can be expected to significantly alter the absorption of the trial drug (e.g. major gastrointestinal tract surgery or inflammatory bowel disease)
* Recent (within 30 days or 5-half-lives, whichever is longer) or current participation in another clinical study in which an investigational medicinal product or device has been received
* Any medical condition or history thereof or any deviation from normal laboratory values that, in the opinion of the investigator, clinically contraindicates or hinders the completion of the trial
* Any reason for suspecting a considerable lack of compliance to the trial

Inclusion criteria for the control group (cross-sectional study alone):

* Age ≥ 40 and ≤ 75 years
* eGFR ≥60ml/min/1,73m2 at screening
* Ability to communicate with the investigator and give informed consent

Exclusion criteria for the control group (cross-sectional study alone):

* Any major chronic disease, e.g. diabetes mellitus, chronic kidney disease, ischemic heart disease, chronic obstructive pulmonary disease (this criterium does not include conditions that may be considered risk factors for chronic diseases, e.g. essential hypertension, primary hypercholesterolemia)
* Acute kidney disease within 3 months
* History of persistent UACR ≥ 30mg/g (in more than two out of three valid measurements over a minimum of three months including those at screening) or a previous diagnosis of micro- or macroalbuminuria
* Current or recent (within 3 months) treatment with ezetimibe
* Any contraindication to an MR-examination (e.g. magnetic foreign body that cannot easily be removed from the body prior to the examination or claustrophobia)
* Any previous major organ transplantation
* Elective major surgery during the study
* Pregnancy, planned pregnancy or breastfeeding during the study
* Severe alcohol consumption or abuse of recreational drugs
* Moderate to severe liver failure (Child Pugh 7-15)
* Recent (within 30 days or 5-half-lives, whichever is longer) or current participation in another clinical study in which an investigational medicinal product or device has been received
* Any medical condition or history thereof or any deviation from normal laboratory values that, in the opinion of the investigator, clinically contraindicates or hinders the completion of the study
* Any reason for suspecting a considerable lack of compliance to the study

Inclusion criteria for the group of participants with T2D and no DKD (cross-sectional study alone):

* Age ≥ 40 and ≤ 75 years
* T2D (World Health Organization criteria)
* eGFR ≥60ml/min/1,73m2 at screening
* Ability to communicate with the Investigator and give informed consent

Exclusion criteria for the group of participants with T2D and no DKD (cross-sectional study alone):

* Any chronic kidney disease
* Acute kidney disease within 3 months
* History of persistent UACR ≥ 30mg/g (in more than two out of three valid measurements over a minimum of three months including those at screening) or a previous diagnosis of micro- or macroalbuminuria
* Current or recent (within 3 months) treatment with ezetimibe
* Any contraindication to an MR-examination (e.g. magnetic foreign body that cannot easily be removed from the body prior to the examination or claustrophobia)
* Any previous major organ transplantation
* Elective major surgery during the study
* Pregnancy, planned pregnancy or breastfeeding during the study
* Severe alcohol consumption or abuse of recreational drugs
* Moderate to severe liver failure (Child Pugh 7-15)
* Recent (within 30 days or 5-half-lives, whichever is longer) or current participation in another clinical study in which an investigational medicinal product or device has been received
* Any medical condition or history thereof or any deviation from normal laboratory values that, in the opinion of the investigator, clinically contraindicates or hinders the completion of the study procedures
* Any reason for suspecting a considerable lack of compliance to the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Urinary albumin creatinine ratio (UACR) | Change over 16 weeks of treatment

SECONDARY OUTCOMES:
Magnetic resonans estimate of kidney parenchymal triglyceride fraction | Change over 16 weeks of treatment

OTHER OUTCOMES:
Urine metabolomic profile | Change over 16 weeks of treatment
  Metabolomic profiling of polar and non-polar urinary metabolites
Plasma extracellular vesicles | Change over 16 weeks of treatment
  number, number from relevant cell types and for all extracellular vesicles the presence of fatty acid transporter proteins
Urine extracellular vesicles | Change over 16 weeks of treatment
  number, number from relevant cell types and for all extracellular vesicles the presence of fatty acid transporter proteins

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided